CLINICAL TRIAL: NCT06053567
Title: Efficacy and Implementation of Exercise-based Smoking Cessation Treatment for Adults With High Anxiety Sensitivity.
Brief Title: Community-based Smoking Cessation Treatment for Adults With High Stress Sensitivity.
Acronym: STEP3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jasper A. Smits (Other)
Collaborators: University of Houston (Other); University of Oklahoma (Other); National Cancer Institute (NCI) (NIH); YMCA (Other)
Responsible Party: Sponsor-Investigator, Jasper A. Smits, Principal Investigator, University of Texas at Austin
Organization: University of Texas at Austin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016120049; R01CA273221 (NIH)
Record Dates: First submitted 2023-09-07; First posted 2023-09-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Exercise; Counseling; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Intensity Aerobic Exercise (Experimental): Participants assigned to this arm will be instructed to complete 75 minutes per week of aerobic training at 60-85% of the their heart rate reserve.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Counseling; Drug: Nicotine patch
- Low-Intensity Aerobic Exercise (Active Comparator): Participants assigned to this arm will be instructed to complete 75 minutes per week of aerobic training at 20-40% of the their heart rate reserve.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Counseling; Drug: Nicotine patch

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants will select a YMCA branch and will be assigned a personal fitness instructor who will oversee a 15-week exercise intervention. The weekly exercise prescription is 75 minutes of aerobic training.
Behavioral: Counseling — Participants will receive the standard tobacco cessation package of up to 5 proactive interactions from the Texas Tobacco Quitline (TTQ). Interactions are typically phone calls, but can be chat or live text if the participant prefers. Interaction 1 is for assessment and quit date planning, Interaction 2 occurs prior to the quit date and can be a group session, Interaction 3 occurs shortly following the quit date, and Interactions 4 and 5 are for relapse prevention if the smoker has quit or problem solving if they have not quit. TTQ also offers a tobacco cessation text messaging program and access to a web portal with a variety of cessation resources.
Drug: Nicotine patch — On the target quit day (week 6), participants will be provided 8 weeks of nicotine replacement therapy (24-hour transdermal nicotine patches [TNP]).

SUMMARY:
Anxiety sensitivity, reflecting the fear of bodily sensations, is a risk factor for the maintenance and relapse of smoking. This study is designed to address the question - is a smoking cessation intervention personalized to high anxiety sensitive smokers and adapted for implementation by the YMCA effective among racially/ethnically diverse samples?

DETAILED DESCRIPTION:
This protocol provides the recommended treatment to achieve smoking cessation (i.e., counseling and nicotine replacement therapy) and randomly assigns individuals to a high-intensity exercise or low-intensity exercise intervention as a strategy to engage the mechanisms relevant to high anxiety sensitive smokers to improve smoking cessation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18);
* High Anxiety Sensitivity (≥5 on the Short Scale Anxiety Sensitivity Index [SSASI]);
* Daily smoker, ≥5 cigarettes (including e-cigarettes, little cigars/cigarillos) for ≥1 year;
* Motivated to quit smoking as evidenced by a score of ≥5 on a 0-10 Likert scale;
* Body mass index <40;
* Medical clearance to participate.
* Located near a participating YMCA site (within 50 miles)

Exclusion Criteria:

* Regular exercise defined as engaging in vigorous-intensity exercise for at least 75 minutes per week for the last 3 months
* Receiving current intervention for smoking cessation.
* Outstanding debt to the YMCA
* Listed as a sex offender on the National Sex Offender Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence abstinence (PPA) at 6-month follow-up | Protocol week 30, which is 24 weeks (6 months) after the quit attempt (set at week 6)
  Self-report of no smoking (not even a puff) during the previous 7 days, verified by expired carbon monoxide (CO; ≤5ppm), saliva cotinine (<30 ng/mL), or significant other, and not invalidated by any of these verification measures. Failure to provide any of these 3 verification measures will result in PPA being considered missing.

SECONDARY OUTCOMES:
7-day point prevalence abstinence (PPA) at 12-month follow-up | Protocol week 54, which is 48 weeks (12 months) after the quit attempt (set at week 6)
  Self-report of no smoking (not even a puff) during the previous 7 days, verified by expired carbon monoxide (CO; ≤5ppm), saliva cotinine (<30 ng/mL), or significant other, and not invalidated by any of these verification measures. Failure to provide any of these 3 verification measures will result in PPA being considered missing.
7-day point prevalence abstinence (PPA) at 9-month follow-up | Protocol week 42, which is 36 weeks (9 months) after the quit attempt (set at week 6)
  Self-report of no smoking (not even a puff) during the previous 7 days, verified by expired carbon monoxide (CO; ≤5ppm), saliva cotinine (<30 ng/mL), or significant other, and not invalidated by any of these verification measures. Failure to provide any of these 3 verification measures will result in PPA being considered missing.

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Smits, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Within one year of completion (publication) of the primary aims for this project, we will provide de-identified data from this project to interested researchers. The data are to be provided in a SPSS file or Excel, with separate documentation of labels/characteristics for each column of data. Data will be released directly by Dr. Smits's team at UT to investigators providing evidence of their institution's IRB approval for planned analyses of the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one year of completion (publication) of the primary aims. No end date.
Access Criteria: Data will be released directly by Dr. Smits's team at UT to investigators providing evidence of their institution's IRB approval for planned analyses of the data.